CLINICAL TRIAL: NCT00607412
Title: AUDs and PTSD Treatment for Victims of Partner Violence
Brief Title: Alcohol Use Disorders (AUDs) and Post-traumatic Stress Disorder (PTSD) Treatment for Victims of Partner Violence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Sonya Norman, PhD, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23AA015707 (NIH); K23AA015707 (NIH)
Record Dates: First submitted 2007-12-26; First posted 2008-02-05 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2009-06

CONDITIONS: PTSD; Substance Use Disorders
Keywords: PTSD; substance use disorders; psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Present focused, integrated psychotherapy for PTSD and substance use disorders
  Interventions: Behavioral: Integrated psychotherapy for PTSD and substance use
- 2 (Active Comparator): Supportive therapy using 12-step model
  Interventions: Behavioral: 12-step based supportive therapy

INTERVENTIONS:
Behavioral: Integrated psychotherapy for PTSD and substance use — integrated, present focused psychotherapy for PTSD and substance use disorders tailored to women who have experienced intimate partner violence
  Arms: 1
Behavioral: 12-step based supportive therapy — supportive psychotherapy based on 12-step model
  Arms: 2

SUMMARY:
The goal of this study is to evaluate a psychotherapy for PTSD and substance use disorders among women who have experienced domestic violence. The hypothesis is that women who receive present-focused, integrated treatment will have greater PTSD symptom reduction and have less substance use after treatment than women in the control condition who will receive supportive therapy based on a 12-step approach.

DETAILED DESCRIPTION:
The goal of this study is to evaluate an integrated psychotherapy for PTSD and substance use disorders among female victims of intimate partner violence. The hypothesis is that women who receive present-focused, integrated treatment will have greater PTSD symptom reduction and have less substance use post-treatment than women in the control condition who will receive supportive therapy based on a 12-step approach.

ELIGIBILITY:
Inclusion Criteria:

* female victims of partner violence
* at least one month out of the abusive relationship
* meet DSM-IV (American Psychiatric Association, 1994) criteria for PTSD and an alcohol use disorder
* literate in English
* have not changed psychotropic medications or dosages within the past two months and agree not to during the active phase (first 12 weeks) of the intervention
* have an identified primary care physician

Exclusion Criteria:

* moderate or severe cognitive impairment as measured by a Mini-Mental State Examination score less than or equal to 18
* Histories of psychosis or mania may be excluded because the presence of these disorders is thought to impede progress in psychotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
CAPS for PTSD symptoms and ASI for substance use | pre, mid treatment, post, 3-month follow-up, 6-month follow-up

SECONDARY OUTCOMES:
Timeline Follow-back procedure, Beck Depression Inventory | same as primary

CONTACTS AND LOCATIONS:
Overall Officials: Sonya Norman, Principal Investigator — UCSD
Locations (1):
- UCSD Outpatient Psychiatry, San Diego, California, United States

REFERENCES:
- [Derived] Hameed M, O'Doherty L, Gilchrist G, Tirado-Munoz J, Taft A, Chondros P, Feder G, Tan M, Hegarty K. Psychological therapies for women who experience intimate partner violence. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD013017. doi: 10.1002/14651858.CD013017.pub2. PMID 32608505
- [Derived] Myers US, Browne KC, Norman SB. Treatment Engagement: Female Survivors of Intimate Partner Violence in Treatment for PTSD and Alcohol Use Disorder. J Dual Diagn. 2015;11(3-4):238-47. doi: 10.1080/15504263.2015.1113762. PMID 26515712